CLINICAL TRIAL: NCT00507442
Title: Phase 1/2 Study of VELCADE® (Bortezomib), Dexamethasone, and Revlimid® (Lenalidomide) Versus VELCADE, Dexamethasone, Cyclophosphamide, and Revlimid Versus VELCADE, Dexamethasone and Cyclophosphamide in Subjects With Previously Untreated Multiple Myeloma
Brief Title: Phase 1/2 Study of VELCADE® in Combination With Other Drugs to Treat Previously Untreated Multiple Myeloma Patients
Acronym: EVOLUTION
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C05008
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Results first posted 2011-12-29 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2012-04

CONDITIONS: Multiple Myeloma
Keywords: Treatment for patients with multiple myeloma; who have received no prior treatment
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Cyclophosphamide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- VDR (Experimental): VELCADE (bortezomib), dexamethasone, and Revlimid (lenalidomide)
  Interventions: Drug: VELCADE (bortezomib); Drug: dexamethasone; Drug: Revlimid (lenalidomide)
- VDCR (Experimental): VELCADE (bortezomib), dexamethasone, cyclophosphamide, Revlimid (lenalidomide)
  Interventions: Drug: VELCADE (bortezomib); Drug: dexamethasone; Drug: cyclophosphamide; Drug: Revlimid (lenalidomide)
- VDC (Experimental): VELCADE (bortezomib), dexamethasone, cyclophosphamide
  Interventions: Drug: VELCADE (bortezomib); Drug: dexamethasone; Drug: cyclophosphamide
- VDC-mod (Experimental): Modified dosing of VELCADE (bortezomib), dexamethasone, cyclophosphamide
  Interventions: Drug: VELCADE (bortezomib); Drug: dexamethasone; Drug: cyclophosphamide

INTERVENTIONS:
Drug: VELCADE (bortezomib) — bortezomib 1.3 mg/m^2 given via IV on days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles, then on days 1, 8, 15 and 22 of a 6-week cycle for 4 cycles (maintenance).
Drug: dexamethasone — dexamethasone 40 mg orally on days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop
Drug: cyclophosphamide — cyclophosphamide 500 mg/m^2 orally on days 1 and 8 of a 3-week cycle for 8 cycles, then stop
  Arms: VDC; VDC-mod; VDCR
Drug: Revlimid (lenalidomide) — lenalidomide 25 mg orally on days 1 to 14 of a 3-week cycle for 8 cycles then stop (VDR arm)
  lenalidomide 15 mg orally on days 1 to 14 of a 3-week cycle for 8 cycles then stop (VDCR arm)
  Arms: VDCR; VDR

SUMMARY:
The purpose of this Phase 1/2 study is to evaluate the efficacy and safety of treatment with VELCADE, dexamethasone, and Revlimid® (VDR) as well as VELCADE, dexamethasone, cyclophosphamide, and Revlimid (VDCR) in patients with multiple myeloma who have received no prior treatment. This study will evaluate whether the addition of Revlimid to VELCADE and Dexamethasone will increase the complete response (CR)/ very good partial response (VGPR) rate.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Male or female subject 18 years of age or older
* A Karnofsky Performance Status score of ≥50% (Eastern Cooperative Oncology Group Performance Status score ≤2)
* Subjects must have symptomatic myeloma or asymptomatic myeloma with myeloma-related organ damage
* Diagnosed Multiple myeloma
* Subjects must have measurable disease requiring systemic therapy
* Subjects must not have been treated previously with any systemic therapy for multiple myeloma
* Two weeks must have elapsed since the date of the last radiotherapy treatment
* Women of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 to 14 days prior to therapy and repeated within 24 hours before starting study drug. They must commit to continued abstinence from heterosexual intercourse or begin 2 acceptable methods of birth control (1 highly effective method and 1 additional effective method) used at the same time, beginning at least 4 weeks before initiation of Revlimid treatment. Women must also agree to ongoing pregnancy testing
* Men must agree to not father a child and agree to use a latex condom during therapy and for 4 weeks after the last dose of study drug, even if they have had a successful vasectomy, if their partner is of childbearing potential
* All subjects must agree to comply with the requirements of the RevAssistSM program

Exclusion Criteria:

* History of allergy to any of the study medications, their analogues, or excipients in the various formulations
* ≥Grade 2 peripheral neuropathy on clinical examination
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or clinically significant conduction system abnormalities.
* Female subject who is pregnant or breast-feeding
* Clinically relevant active infection or serious comorbid medical conditions
* Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he/she were to participate in the study. This includes but is not limited to serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Active prior malignancy diagnosed or treated within the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Kumar S, Flinn I, Richardson PG, Hari P, Callander N, Noga SJ, Stewart AK, Turturro F, Rifkin R, Wolf J, Estevam J, Mulligan G, Shi H, Webb IJ, Rajkumar SV. Randomized, multicenter, phase 2 study (EVOLUTION) of combinations of bortezomib, dexamethasone, cyclophosphamide, and lenalidomide in previously untreated multiple myeloma. Blood. 2012 May 10;119(19):4375-82. doi: 10.1182/blood-2011-11-395749. Epub 2012 Mar 15. PMID 22422823
- [Derived] Kumar SK, Flinn I, Noga SJ, Hari P, Rifkin R, Callander N, Bhandari M, Wolf JL, Gasparetto C, Krishnan A, Grosman D, Glass J, Sahovic EA, Shi H, Webb IJ, Richardson PG, Rajkumar SV. Bortezomib, dexamethasone, cyclophosphamide and lenalidomide combination for newly diagnosed multiple myeloma: phase 1 results from the multicenter EVOLUTION study. Leukemia. 2010 Jul;24(7):1350-6. doi: 10.1038/leu.2010.116. Epub 2010 May 27. PMID 20508619

RESULTS

PARTICIPANT FLOW:
Groups:
- V-DR: VELCADE (bortezomib), dexamethasone, and Revlimid (lenalidomide) Bortezomib: 1.3 mg/m^2/dose IV on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles, then on Days 1, 8, 15, and 22 of a 6-week cycle for 4 cycles.
  Dexamethasone: 40 mg orally [PO] on Days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop.
  Lenalidomide: 25 mg PO on Days 1 through 14 of a 3-week cycle for 8 cycles, then stop.
- VDCR: VELCADE (bortezomib), dexamethasone, cyclophosphamide, Revlimid (lenalidomide) Bortezomib: 1.3 mg/m^2/dose IV on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles, then on Days 1, 8, 15, and 22 of a 6-week cycle for 4 cycles.
  Dexamethasone: 40 mg PO on Days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop.
  Cyclophosphamide: 100 - 500 mg/m^2 dose PO on Days 1 and 8 of a 3-week cycle for 8 cycles, then stop.
  Lenalidomide: 15 mg PO on Days 1 through 14 of a 3-week cycle for 8 cycles, then stop.
- V-DC: VELCADE (bortezomib), dexamethasone, cyclophosphamide Bortezomib: 1.3 mg/m^2/dose IV on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles, then on Days 1, 8, 15, and 22 of a 6-week cycle for 4 cycles.
  Dexamethasone: 40 mg orally PO on Days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop.
  Cyclophosphamide: 500 mg/m^2 dose PO on Days 1 and 8 of a 3-week cycle for 8 cycles, then stop.
- VDC-mod: Modified dosing of VELCADE (bortezomib), dexamethasone, cyclophosphamide Bortezomib: 1.3 mg/m^2/dose IV on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles, then on Days 1, 8, 15, and 22 of a 6-week cycle for 4 cycles.
  Dexamethasone: 40 mg PO on Days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop.
  Cyclophosphamide: 500 mg/m^2 dose PO on Days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop.
Period: Overall Study
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Started | 42 | 66 | 33 | 17
Completed | 26 | 39 | 18 | 12
Not Completed | 16 | 27 | 15 | 5
Not completed — Adverse Event | 8 | 11 | 4 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 4 | 1
Not completed — Progressive Disease | 2 | 4 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 2 | 1
Not completed — Other | 2 | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V-DR | VDCR | V-DC | VDC-mod | Total
Number analyzed (Participants) | 42 | 66 | 33 | 17 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 42 | 21 | 11 | 101
  >=65 years | 15 | 24 | 12 | 6 | 57
Age Continuous [Mean (Standard Deviation); unit: years] | 59.5 (8.76) | 60.9 (8.97) | 61.4 (8.32) | 59.6 (9.16) | 60.5 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 28 | 14 | 10 | 70
  Male | 24 | 38 | 19 | 7 | 88
Region of Enrollment [Number; unit: participants]
  United States | 42 | 66 | 33 | 17 | 158

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Combined Complete Response and Very Good Partial Response
Description: Complete response requires negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow.
  Very good partial response requires serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 h
Time Frame: Up to 48 weeks or until disease progression
Population: The response-evaluable population is defined as phase 2 patients with measurable disease at baseline and with at least 1 post baseline response assessment.
Measure: Number; unit: participants
Groups:
- V-DR: Bortezomib: 1.3 mg/m^2/dose IV on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles, then on Days 1, 8, 15, and 22 of a 6-week cycle for 4 cycles.
  Dexamethasone: 40 mg orally [PO] on Days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop.
  Lenalidomide: 25 mg PO on Days 1 through 14 of a 3-week cycle for 8 cycles, then stop.
- VDCR: Bortezomib: 1.3 mg/m^2/dose IV on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles, then on Days 1, 8, 15, and 22 of a 6-week cycle for 4 cycles.
  Dexamethasone: 40 mg PO on Days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop.
  Cyclophosphamide: 500 mg/m^2 dose PO on Days 1 and 8 of a 3-week cycle for 8 cycles, then stop.
  Lenalidomide: 15 mg PO on Days 1 through 14 of a 3-week cycle for 8 cycles, then stop.
- V-DC: Bortezomib: 1.3 mg/m^2/dose IV on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles, then on Days 1, 8, 15, and 22 of a 6-week cycle for 4 cycles.
  Dexamethasone: 40 mg orally PO on Days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop.
  Cyclophosphamide: 500 mg/m^2 dose PO on Days 1 and 8 of a 3-week cycle for 8 cycles, then stop.
- VDC-mod: Bortezomib: 1.3 mg/m^2/dose IV on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles, then on Days 1, 8, 15, and 22 of a 6-week cycle for 4 cycles.
  Dexamethasone: 40 mg PO on Days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop.
  Cyclophosphamide: 500 mg/m^2 dose PO on Days 1, 8, and 15 of a 3-week cycle for 8 cycles, then stop.
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 41 | 40 | 32 | 17
participants | 21 | 23 | 13 | 9

2. Secondary Outcome: Number of Patients With Adverse Events (AEs)
Description: Evaluate the safety and tolerability of the combination therapy
Time Frame: From first dose of study drug through the 30 day post-treatment AE assessment visit
Population: The safety population includes patients received any dose of any study drug.
Measure: Number; unit: participants
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 42 | 66 | 33 | 17
participants | 42 | 65 | 33 | 17

3. Secondary Outcome: Number of Patients With Overall Response
Description: Overall Response includes complete response and partial response.
  Complete response requires negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow.
  Partial response requires at least 50% reduction of serum M-protein and reduction in 24-h urinary M-protein by at least 90% or to < 200 mg per 24 hour.
Time Frame: Up to 48 weeks or until disease progression
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 41 | 40 | 32 | 17
participants | 35 | 35 | 24 | 17

4. Secondary Outcome: Number of Patients With Stringent Complete Response Rate
Description: Stringent Complete Response is defined as complete response plus normal free light chain (kappa/lambda) ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence.
Time Frame: Up to 48 weeks or until disease progression
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 41 | 40 | 32 | 17
participants | 7 | 6 | 3 | 5

5. Secondary Outcome: Number of Patients With Complete Response Rate + Near Complete Response Rate
Description: Complete response requires negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow.
  Near Complete response requires positive immunofixation on the serum and/or urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow.
Time Frame: Up to 48 weeks or until disease progression
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 41 | 40 | 32 | 17
participants | 17 | 14 | 10 | 8

6. Secondary Outcome: Duration of Response
Description: Duration of response is the time from date of first documented confirmed response to date of first documented progressive disease. A confirmed response is a response that has been observed on at least two consecutive assessments.
  Disease progression requires any one or more of the following: serum m-protein increase >= 25% from nadir(absolute increase >= 0.5 g/dL); Urine m-protein increase >= 25% from nadir(absolute increase >= 200 mg/24 hr), bone marrow plasma cell percentage increase >= 25% from nadir(absolute increase >= 10%), new bone lesion or soft tissue plasmacytomas.
Time Frame: Up to 48 weeks or until disease progression
Population: Responders (patients achieved complete and partial response) in the response evaluable population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 35 | 35 | 24 | 17
days | NA [302 to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [583 to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [NA to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [NA to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time

7. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as time from the date of randomization to the date of first documented progressive disease.
  Disease progression requires any one or more of the following: serum m-protein increase >= 25% from nadir(absolute increase >= 0.5 g/dL); Urine m-protein increase >= 25% from nadir(absolute increase >= 200 mg/24 hr), bone marrow plasma cell percentage increase >= 25% from nadir(absolute increase >= 10%), new bone lesion or soft tissue plasmacytomas.
Time Frame: Up to 48 weeks or until disease progression
Population: The modified intent-to-treat population is defined as phase 2 patients received at least one dose of any drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 42 | 48 | 33 | 17
days | NA [NA to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [631 to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [NA to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [NA to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time

8. Secondary Outcome: Time to Response
Description: Time to response is defined as time from date of randomization to the date of the first documentation of a confirmed response. confirmed response is a response that has been observed on at least two consecutive assessments.
Time Frame: Up to 48 weeks or until disease response
Population: Responders (patients achieved complete and partial response) in the response evaluable population.
Measure: Median (Full Range); unit: days
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 35 | 35 | 24 | 17
days | 49 [43 to 175] | 50 [41 to 145] | 55 [42 to 302] | 49 [42 to 194]

9. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as time from the date of randomization to the date of the first documented progressive disease or death.
  Disease progression requires any one or more of the following: serum m-protein increase >= 25% from nadir(absolute increase >= 0.5 g/dL); Urine m-protein increase >= 25% from nadir(absolute increase >= 200 mg/24 hr), bone marrow plasma cell percentage increase >= 25% from nadir(absolute increase >= 10%), new bone lesion or soft tissue plasmacytomas.
Time Frame: Up to 48 weeks or until disease progression/death
Population: The modified intent-to-treat population is defined as phase 2 patients received at least one dose of any drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 42 | 48 | 33 | 17
days | NA [356 to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | 631 [555 to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [778 to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [NA to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time

10. Secondary Outcome: Probability of 1-year Survival
Time Frame: survival probability at 1 year after randomization
Population: The modified intent-to-treat population is defined as phase 2 patients received at least one dose of any drug.
Measure: Number; unit: percentage of patients
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 42 | 48 | 33 | 17
percentage of patients | 100 | 91.6 | 100 | 100

11. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from the date of randomization to the date of death
Time Frame: Up to 48 weeks or until death
Population: The modified intent-to-treat population is defined as phase 2 patients received at least one dose of any drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Number analyzed (Participants) | 42 | 48 | 33 | 17
days | NA [NA to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [NA to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [NA to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time | NA [NA to NA] — Not estimable based on the Kaplan-Meier method because of insufficient follow up time

ADVERSE EVENTS:
Time Frame: From first dose of any study drug to 30-day post-treatment adverse event assessment, up to 48 weeks and 30 days
Description: From first dose of any study drug to end of treatment period
Arm/Group | V-DR | VDCR | V-DC | VDC-mod
Serious Adverse Events (participants affected / at risk) | 17/42 | 26/66 | 7/33 | 7/17
Other Adverse Events (participants affected / at risk) | 41/42 | 65/66 | 33/33 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V-DR (N=42) | VDCR (N=66) | V-DC (N=33) | VDC-mod (N=17)
Pneumonia NOS (Infections and infestations) | 2 | 3 | 0 | 1
Lobar pneumonia NOS (Infections and infestations) | 1 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection NOS (Infections and infestations) | 0 | 0 | 2 | 0
Respiratory syncytial virus infection NOS (Infections and infestations) | 0 | 1 | 0 | 0
Arthritis infective NOS (Infections and infestations) | 0 | 0 | 1 | 0
Colitis pseudomembranous (Infections and infestations) | 1 | 0 | 0 | 0
Stye (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection NOS (Infections and infestations) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 1 | 3 | 1 | 0
Small intestinal obstruction NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diverticular perforation NOS (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea NOS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Antibiotic associated colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Weakness (General disorders) | 0 | 0 | 0 | 1
Fall (General disorders) | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Neuralgia NOS (General disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 5 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Malnutrition NOS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain aggravated (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hypotension NOS (Vascular disorders) | 1 | 2 | 2 | 0
Venous thrombosis deep limb (Vascular disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Pulmonary oedema NOS (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis NOS (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Renal failure NOS (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal impairment NOS (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 2
Headache NOS (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsions NOS (Nervous system disorders) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0
Blood culture positive (Investigations) | 0 | 1 | 0 | 0
Haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle injury NOS (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Hypoproteinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Caecitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anaemia NOS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia NOS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | V-DR (N=42) | VDCR (N=66) | V-DC (N=33) | VDC-mod (N=17)
Peripheral neuropathy NOS (Nervous system disorders) | 14 | 24 | 15 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 17 | 26 | 9 | 1
Dizziness (excl vertigo) (Nervous system disorders) | 13 | 18 | 4 | 3
Dysgeusia (Nervous system disorders) | 8 | 9 | 3 | 1
Paraesthesia (Nervous system disorders) | 4 | 6 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 5 | 4 | 0
Tremor (Nervous system disorders) | 5 | 5 | 1 | 1
Constipation (Gastrointestinal disorders) | 26 | 29 | 16 | 7
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 2 | 6 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 6 | 8 | 3
Abdominal distension (Gastrointestinal disorders) | 8 | 3 | 1 | 4
Flatulence (Gastrointestinal disorders) | 2 | 4 | 1 | 1
Hiccups (Gastrointestinal disorders) | 3 | 6 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 6 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 3 | 2 | 0
Pharyngolaryngeal pain (Gastrointestinal disorders) | 3 | 6 | 1 | 2
Oedema lower limb (General disorders) | 9 | 19 | 8 | 5
Rigors (General disorders) | 11 | 14 | 5 | 2
Pain NOS (General disorders) | 6 | 7 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 7 | 7 | 4 | 0
Pruritus NOS (Skin and subcutaneous tissue disorders) | 5 | 6 | 2 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 5 | 1 | 2
Sweating increased (Skin and subcutaneous tissue disorders) | 3 | 7 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 5 | 9 | 2 | 1
Rash NOS (Skin and subcutaneous tissue disorders) | 1 | 6 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 1
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 3
Pain in limb (Musculoskeletal and connective tissue disorders) | 12 | 22 | 12 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 14 | 5 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 3 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1 | 1
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 5 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 8 | 33 | 17 | 8
Lymphopenia (Blood and lymphatic system disorders) | 5 | 6 | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 15 | 5 | 2
Appetite decreased NOS (Metabolism and nutrition disorders) | 6 | 5 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 8 | 4 | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 6 | 4 | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 4 | 2 | 2
Insomnia (Psychiatric disorders) | 14 | 21 | 9 | 6
Anxiety NEC (Psychiatric disorders) | 4 | 10 | 1 | 1
Depression NOS (Psychiatric disorders) | 1 | 7 | 1 | 1
Weight decreased (Investigations) | 3 | 5 | 6 | 1
Weight increased (Psychiatric disorders) | 1 | 3 | 4 | 1
Alanine aminotransferase increased (Investigations) | 4 | 1 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 3 | 2
Haemoglobin decreased (Investigations) | 1 | 2 | 4 | 3
Nasopharyngitis (Infections and infestations) | 4 | 8 | 4 | 2
Vision blurred (Eye disorders) | 7 | 6 | 4 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 3 | 2 | 2
Muscle cramps (Musculoskeletal and connective tissue disorders) | 7 | 9 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 1 | 1
Day mouth (Gastrointestinal disorders) | 3 | 4 | 0 | 1
Flushing (Vascular disorders) | 2 | 5 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No